CLINICAL TRIAL: NCT06046404
Title: Refraining From Closed Reduction of Dislocated Distal Radius Fractures in the Emergency Department
Acronym: RECORDED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L2022093
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-09

CONDITIONS: Wrist Fractures; Distal Radius Fractures; Closed Reduction of Fracture and Application of Plaster Cast; Wrist Injuries; Radius Fracture Distal
MeSH Terms: conditions — Wrist Fractures; Wrist Injuries | interventions — Closed Fracture Reduction

STUDY DESIGN:
Masking Description: cluster randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- closed reduction followed by plaster casting (Active Comparator)
  Interventions: Procedure: closed reduction
- only plaster casting (Experimental): no closed reduction will be performed
  Interventions: Procedure: no closed reduction

INTERVENTIONS:
Procedure: closed reduction — the intervention of closed fracture reduction widely known and part of daily practice. we test the eficacy of this intervention by not performing it in our test group.
  Arms: closed reduction followed by plaster casting
Procedure: no closed reduction — no reduction will be performed
  Arms: only plaster casting

SUMMARY:
The investigators test the efficacy of closed reduction in displaced distal radial fractures in the emergency department.

DETAILED DESCRIPTION:
in a multicenter cluster randomized trial the investigators aim to include 134 patients with displaced distal radial fractures awaiting surgery and randomize between closed reduction followed by plaster casting and plaster casting alone. Primairy outcomes are pain in the days leading up to surgery and postoperative hand- and wrist function. Secondary outcomes are length of stay in the emergency department, length of surgey, return to work and complications.

ELIGIBILITY:
Inclusion Criteria:

* displaced distal radial fracture eligible for surgery

Exclusion Criteria:

* ISS traumascore >16
* open fracture
* multiple fractures in ipsilateral extremety
* neurovascular damage
* previous injury in the same wrist
* inability to complete questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
daily pain scores | usually 2-10 days
  pain reported in the days awaiting surgery on the visual analog scale (VAS) scoring from 0 to 10 where 0 equals no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
function | 6 weeks, 3, 6 and 12 months
  hand function as reported by the patient reported hand and wrist evaluation (PRHWE) questionnaire. scoring from 0 to 100 with 0 meaning perfect function with no impairment or pain and 100 meaning no function at all with maximum pain.
Number of complications | 1 year
  The investigators will report all complications including, but not limited to: nerve damage, CRPS, infection, bleeding, malunion and need for revision surgery will be tracked.
Wrist mobility | 6 weeks and 3 months
  Range of motion will be reported in form of wrist flexion and extension and pro- and supination, in degrees.
length of stay in emergency department | baseline
  length of stay in emergency department
quality of life in EQ5D5L | 1 year
  reported by the EQ5D5L questionnaire. EQ-5D-5L health states can be summarised using a 5-digit code or represented by a single summary number (index value), which reflects how good or bad a health state is according to the preferences of the general population of a country/region.

CONTACTS AND LOCATIONS:
Locations (1):
- Maasstad Hospital, Rotterdam, Maasstadweg 21, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided